CLINICAL TRIAL: NCT01406795
Title: Evaluation of GORE VIABAHN Endoprosthesis With Heparin Bioactive Surface for the Treatment of Venous Occlusions and Stenoses
Brief Title: The GORE Viabahn Endoprosthesis for the Treatment of Venous Occlusions and Stenoses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment and advances in venoplasty only techniques of the femoral vein
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lawrence (Rusty) Hofmann, Chief of Interventional Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-01312011-7377; FDA IDE - G090054; IRB eProtocol - 14781; SPO # 49275
Record Dates: First submitted 2011-07-22; First posted 2011-08-01 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Venous Thrombosis
Keywords: Post Thrombotic Syndrome; Venous Stasis; Venous Occlusions; Venous Stenosis
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome; Varicose Ulcer

ARMS (1):
- Venous Stent Arm (Experimental): The study is a single treatment arm study and the venous stent will be placed in all eligible participants.
  Interventions: Device: Gore Viabahn Heparin Coated Stent

INTERVENTIONS:
Device: Gore Viabahn Heparin Coated Stent — For subjects deemed to be suffering from chronic venous insufficiency of the femoral or popliteal veins, a Gore Viabahn stent will be implanted during a venoplasty procedure to determine whether the vein will stay open.

SUMMARY:
To study the safety and efficacy of drug coated stents for the treatment of venous occlusions and stenoses in the lower extremity. The use of the device for the treatment of peripheral arterial disease is approved by the FDA, however, the use of the device in venous occlusions and stenoses, although performed by some practitioners, has not yet been studied in detail.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* Patient has clinical manifestations (i.e. symptoms and/or signs) of chronic DVT of an extremity. The Venous Clinical Severity Score (VCSS) will be used to determine if the patient is currently suffering from chronic DVT, with a VCSS score of 4 or greater necessary for inclusion.
* Imaging confirmation of venous occlusion or stenosis (>50%) involving the femoral, and/or popliteal veins
* Obstructed vessel caliber can accommodate a 7FR System, from insertion site to target segment
* Patient is able to read and answer a questionnaire in English

Exclusion Criteria:

* History of life-threatening reaction to contrast material
* Unwilling or unable to provide informed consent, or return for required follow-up evaluations
* Participating in another investigational study that has not completed follow-up testing
* Cannot receive outpatient anticoagulation such as LMWH and/or vitamin K antagonists (VKAs)
* Absolute contraindication to contrast media or renal insufficiency (baseline creatinine >2.0 mg/dL).
* Either a history or presence of heparin-induced thrombocytopenia antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lawrence (Rusty) Hofmann MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited a single patient in 2012 at the Stanford Medical Center. The study ended in 2013.
Period: Overall Study
Arm/Group | Venous Stent Arm
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Stent Migration
Description: Stent migration is reported as the count of participants with stent migration within 1 month following stent placement.
Time Frame: up to 1 month following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: Stent Migration
Description: Stent migration is reported as the count of participants with stent migration within 1 year following stent placement.
Time Frame: up to one year following the procedure 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Participants | 0

3. Primary Outcome: Primary Patency Rate
Description: Patency refers to whether the stent is unoccluded (open). Primary patency rate was defined as the count of participants with >= 50% patency following initial stent placement, and is reported as the count of participants meeting this criteria.
Time Frame: up to 1 year following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Freedom From Device-related Amputation
Description: Freedom from device-related amputation (amputation of infected limb) is reported as the count of participants with no device-related amputation within 1 year following stent placement.
Time Frame: up to 1 year following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Assisted-primary Patency
Description: Patency refers to whether the stent is unoccluded (open). Primary refers to the first time a stent was placed (or the first time patency needed to be established). Assisted refers to the fact that a device (like a balloon) was used to open the stent. Assisted-primary patency is defined as the count of participants that demonstrated the need for an intervention to establish patency.
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Secondary Patency
Description: Secondary patency means that the initial intervention failed and a second intervention was performed to establish or maintain patency. Secondary patency is defined as the count of participants that required a second intervention to establish patency.
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Participants | 0

7. Secondary Outcome: Adverse Events
Description: Adverse events were reported as the count of participants that experienced an adverse event within two years of their procedure.
Time Frame: up to two years 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Participants | 0

8. Secondary Outcome: Decrease in Swelling of Affected Extremity
Description: The count of participants that experienced a decrease in swelling after the stent was placed.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Participants | 0

9. Secondary Outcome: Venous Clinical Severity Score
Description: Venous Clinical Severity represents the severity of the venous pathology, which includes measures like pain, inflammation, and number of ulcers. It is scored on a scale of 0-3 with the upper end representing very severe outcomes for the patient.
Time Frame: up to 2 years
Population: Data were not collected for this outcome
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 0

10. Secondary Outcome: VEINS-QOL
Description: The VEINS-QOL is a questionnaire that represents a patient's quality of life, using measures like how well the patient can walk, sleep, and enjoy life. Responses are graded on a scale of 1-5, with 1 being very good, and 5 being very poor. The VEINS-QOL measure is defined by the count of participants that showed a decreased overall score following their procedure.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 1
Participants | 1

11. Secondary Outcome: Villalta PTS Scale
Description: The Villalta PTS Scale is a score based on the patient's symptoms, includes cramps, pain, and redness. It is scaled from 0 to 48, with a higher score representing more severe disease.
Time Frame: up to 2 years
Population: Data were not collected for this outcome.
Arm/Group | Venous Stent Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Venous Stent Arm
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was underpowered, enrolling only a single patient (goal enrollment was 15 patients).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No